CLINICAL TRIAL: NCT04243707
Title: Diagnostics and Therapy of a Cobalamin Deficiency
Brief Title: Cobalamin Deficiency - Diagnosis and Therapy
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01295
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Vitamin B 12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In a retrospective study with existing values of vitamin B12 and holotranscobalamin 4 strategies are simulated and the results and costs are compared.

Generally, cobalamin ist substituted by intramuscular administration. However, oral preparations are also available. Aims of the focus groups are to investigate the awareness of a (potential) deficiency and to identify a therapy for best adherence.

DETAILED DESCRIPTION:
Various diagnostic strategies exist for the identification of a cobalamin deficiency. In a retrospective study with existing serum values of vitamin B12 and holotranscobalamin 4 strategies are simulated and the results and costs are compared.

A cobalamin deficiency can have various causes: Dietary habits (vegetarian, vegan), advanced age, pernicious anaemia, gastrectomy, drug interactions (metformin, proton pump blocker). Therapy is often performed by intramuscular administration of cobalamin. However, oral preparations are also available in very different dosages. Investigators want to investigate with focus groups whether different patient groups are aware of a (potential) deficiency, how cobalamin is actually substituted (with registered or otherwise acquired products) and which therapy would lead to best adherence.

ELIGIBILITY:
Inclusion Criteria:

* potential cobalamin deficiency

Exclusion Criteria:

* refusal to take part in a survey

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: potential cobalamin deficiency
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
diagnostic strategies | 2017 - 2018
  Sensitivity and specificity of 4 different diagnostic strategies compared to the simultaneous determination of vitamin B12 and holotranscobalamin.
supplementation of cobalamin deficiency | 2020
  Patient's awareness of a potential cobalamin deficiency, treatment actually applied - with or without registration, ideal supplementation to achieve best adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Arnet, PD Dr., Principal Investigator — Pharmaceutical Care Research Group
Locations (1):
- Pharmaceutical Care Research Group, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No